CLINICAL TRIAL: NCT06783556
Title: The Analgesia Effect of Electroacupuncture of Battlefield Acupuncture (BFA) Versus Sham Electroacupuncture on Pain, Analgesic Dose Reduction and Quality of Life Post Percutaneous Nephrolithotomy Surgery
Brief Title: The Analgesia Effect of Electroacupuncture Battlefield Acupuncture Versus Sham Electroakupuncture Post Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Hermin Widyaprastuti, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 24-12-1845
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Percutaneous Nephrolithotomy

STUDY DESIGN:
Intervention Model Description: The Ear Electroacupuncture of Battlefield Acupuncture (BFA) and paracetamol intravenous therapy will be designated as the intervention group, while the sham electroacupuncture and paracetamol intravenous therapy will be designated as the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants, the outcome assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): The Ear Electroacupuncture of Battlefield Acupuncture (BFA) and paracetamol intravenous therapy
  Interventions: Device: The Ear Electroacupuncture of Battlefield Acupuncture (BFA) and paracetamol intravenous therapy
- Control Group (Sham Comparator): The sham electroacupuncture and paracetamol intravenous therapy
  Interventions: Device: The sham electroacupuncture and paracetamol intravenous therapy

INTERVENTIONS:
Device: The Ear Electroacupuncture of Battlefield Acupuncture (BFA) and paracetamol intravenous therapy — Electroacupuncture therapy was performed 2 hours before PCNL surgery. Needle insertion was performed perpendicularly at the Battlefield Acupuncture (BFA) points of the ear, namely MA-IT1 Cingulate gyrus, MA-AT2 Thalamus, MA-H2 Omega2, MA-H1 Point Zero and MA-TF1 Shenmen bilaterally. Then the electrostimulator cable was connected to the ear acupuncture points MA-AT2 and MA-TF1 bilaterally on the same side and then fixed with plaster. Electroacupuncture uses continuous waves of 2 Hz frequency with an intensity that can be tolerated by the patient for 30 minutes.
  Patients also received standard therapy with 1000 mg intravenous paracetamol with a maximum of 3 times administration per 24 hours and can be reduced according to the needs of the patient's pain complaints.
  Arms: Intervention Group
Device: The sham electroacupuncture and paracetamol intravenous therapy — Sham electroacupuncture therapy was performed 2 hours before PCNL surgery. Needle only attached using plester (not inserted) at the Battlefield Acupuncture (BFA) points of the ear, namely MA-IT1 Cingulate gyrus, MA-AT2 Thalamus, MA-H2 Omega2, MA-H1 Point Zero and MA-TF1 Shenmen bilaterally. Then the electrostimulator cable was connected to the ear acupuncture points MA-AT2 and MA-TF1 bilaterally on the same side and then fixed with plaster. Electroacupuncture device is not turned on. The therapy is carried out for 30 minutes.
  Patients also received standard therapy with 1000 mg intravenous paracetamol with a maximum of 3 times administration per 24 hours and can be reduced according to the needs of the patient's pain complaints.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn the effect of ear electroacupuncture BFA therapy in reducing pain, analgesic dose, and improving patient quality of live post percutaneous nephrolithotomy surgery. The main questions it aims to answer are:

* Does BFA ear electroacupuncture reduce postoperative pain of percutaneous nephrolithotomy surgery better than sham electroacupuncture group?
* Does BFA ear electroacupuncture reduce postoperative analgesic dose of percutaneous nephrolithotomy surgery better than sham electroacupuncture group?
* Does BFA ear electroacupuncture improve postoperative quality of life of percutaneous nephrolithotomy surgery better than sham electroacupuncture group?

Researchers will compare ear electroacupuncture BFA to sham electroacupuncture to see the different analgesia effect between these groups.

Participants will:

* Get ear electroacupuncture BFA or sham electroacupuncture therapy, 2 hours before surgery for 30 minutes
* Take drug paracetamol 1000 mg intravenous after surgery according to the needs of the patient's pain complaints after surgery in both groups

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-65 years
* Patients who have been diagnosed with kidney stones measuring > 2 cm and will undergo PCNL surgery
* VAS score <7, assessed 2 hours before PCNL surgery
* Receive standard analgesic therapy
* Willing to participate in this study until completion and sign an informed consent.

Exclusion Criteria:

* Kidney anatomical abnormalities
* Ear deformities (microtia)
* Patients with cognitive impairment, uncooperative (receiving antidepressants or strong opioid or narcotic analgesics)
* Tumors, wounds or skin infections in the needling area.
* Heart rhythm disorder, unstable hemodynamics that require intensive care including extremely high body temperature and using a pacemaker.
* Allergy to acupuncture needles or certain metals
* Patients who have had a DJ stent or nephrostomy before PCNL
* History of metal implants in the body except amalgam

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Before therapy, minute 0, hour 8, hour 24, hour 48
  Visual Analogue Scale is the tool that measures pain intensity. It use a scale with a minimum range of 0 and a maximum of 10, where 0 indicates no pain and 10 indicates the worst pain. Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Analgesic dose reduction | hour 8, hour 24, hour 48
  Paracetamol 1000 mg IV is given to patient with a maximum of 3 times administration per 24 hours. The dose of paracetamol can be reduced when the patien's pain score of Visual Analogue Score is less than 3. Measurements were made by measuring the cumulative dose of analgesics after acupuncture therapy. Then compared between the two groups, which group had a greater decrease in analgesic dose.
Short Form 36 (SF-36) Questionnaire | Before therapy, day 7
  The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). To score the SF-36, scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100. Higher scores indicate better health status.
Adverse effects | Day 7
  Record the adverse effects that occur after acupuncture therapy. It will be monitored for 7 days after therapy and recorded on the 7th day by assessor.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No